CLINICAL TRIAL: NCT03980366
Title: Use of Electroconvulsive Therapy to Treat Self-Injurious Behavior in Adults With Autism Spectrum Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have not obtained additional subjects and chose to terminate/close this study.
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Sentara Norfolk General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT4ASD
Record Dates: First submitted 2019-04-11; First posted 2019-06-10 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-07

CONDITIONS: Autism Spectrum Disorder; Self-Injurious Behavior
Keywords: Electroconvulsive Therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Subjects and their legally-appointed guardians will participate in a total of 18 visits over the course of 1 year. Visits 1 and 2 will occur during weeks 1 and 2. These visits will be for psychiatric and medical evaluations and will take about 1 hour each. Visits 3-14 will take place three times a week for four weeks. These visits will be for the ECT treatments and will take about 2-3 hours each. Visit 15 will take place 1 week post-treatment and visit 16 will take place 4 weeks post-treatment. Guardians will keep a daily diary card between visits 1 and 16, spanning a time of 10 weeks. Visits 17 and 18 will take place at 6 months and 12 months, respectively, and take about 1 hour each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECT to treat self-injurious behaviors in adults with ASD (Experimental): After initial exams and pre-screening, participants will receive bilateral Electroconvulsive Therapy (ECT) for 12 treatments sessions over the course of 4 weeks, plus non-ECT follow-up sessions at 1, 2, 6, and 12 months post-ECT treatment.
  Interventions: Device: Electroconvulsive Therapy (ECT)

INTERVENTIONS:
Device: Electroconvulsive Therapy (ECT) — Bilateral Electroconvulsive Therapy (ECT) to treat self-injurious behavior in adults with Autism Spectrum Disorder (ASD).

SUMMARY:
The purpose of this study is to use formal measures to monitor the outcome of using electroconvulsive therapy to treat self-injurious behavior in adults with Autism Spectrum Disorder for whom psychotropic medication has not worked. This study will be fundamentally different from the previously published literature on the subject in that this will be a prospective study which will aim to recruit multiple participants in an open label study.

DETAILED DESCRIPTION:
Potential participants will be screened for inclusion/exclusion criteria. They must have a confirmed ASD diagnosis and be generally healthy. As part of the inclusion and exclusion criteria, the participant must have an appointment with their primary care provider or a hospital internist to complete a physical exam and required tests (EKG, CXR [chest x-ray], CMP [Comprehensive Metabolic Profile], CBC [Complete Blood Count], and head CTscan). At the first pre-treatment appointment (Visit 1), the participant and their legal guardian will review and sign the consent and assent forms with the investigator. The legal guardian also sign a Sentara Norfolk General Hospital release of medical information. The guardian will then fill out the ASD Diagnostic Checklist, Repetitive Behavior Scale- Revised, and the Aberrant Behavior Checklist. The physician will complete the Self-Injury Trauma Scale, which documents the number, type, and severity of unhealed self-injury traumas. At the end of the Visit 1, the guardian will receive a Subject Diary Card to record the number of self-injury episodes per day, the number of aggressive episodes per day, and the perceived severity of episodes that day. The Diary Card also has space to record the medication taken by the participant every day.

The second pre-treatment appointment (Visit 2) will consist of a complete psychiatric evaluation with review of all medical evaluations. The subject must receive medical clearance to undergo ECT treatment. The first Diary Card will be collected at this time, and a second Diary Card will be given.

After receiving medical clearance, participants (accompanied by their guardians) will begin to receive ECT treatments. They will receive ECT 3 times a week for 4 weeks, for a total of 12 treatments (Visits 3- 14). All ECT treatments will take place in the Outpatient Surgery and Diagnostic Unit of Sentara Norfolk General Hospital, and will be performed by Dr. Shriti Patel or Dr. Justin Petri. All subjects will receive bilateral ECT. Participants will be placed under general anesthesia (Etomidate) and given a primary muscle relaxant (Succinylcholine). An anesthesiologist or nurse anesthetist will be present and will hyperventilate the patient to lower their seizure threshold. The first ECT treatment (Visit 3) will determine the participant's seizure threshold. Subsequent ECT treatments (Visits 4-14) will be determined by the acting psychiatrist based on the patient's seizure threshold. Following the procedure, the patient will recover in the Post Anesthesia Care Unit.

Throughout the course of the treatment, guardians will continue filling out the Diary Card. Once treatment begins, guardians will be asked to also include any side effects of the treatment noted by themselves or the participant. Guardians will turn in and receive new Diary Cards weekly.

After acute ECT treatment is complete, patients and their guardians will return to Eastern Virginia Medical School (EVMS) Department of Psychiatry and Behavioral Sciences for post-treatment appointments (Visits 15-18). At these post-treatment appointment guardians will complete the ASD Diagnostic Checklist, Repetitive Behavior Scale- Revised, and the Aberrant Behavior Checklist. The psychiatrist will complete a second Self-Injury Trauma Scale. At this time the Diary Card will be collected and subjects will receive Diary Cards for 1 month. Visits 15-18 will occur at 1 month, 2 months, 6 months, and 12 months post - acute ECT treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must have:

* a documented Autism Spectrum Disorder diagnosis
* a present history of self-injurious behavior for which they have tried and failed at least four other treatment methods
* a legal guardian who is able to consent to medical treatments and attend all appointments with the participant.
* Subjects will obtain an EKG, Chest X-Ray, Complete Metabolic Panel, Complete Blood Count, and a head CT to receive medical clearance prior to participating in the ECT.

Exclusion Criteria:

Participants will be excluded if they are:

* under the age of 18
* older than age of 89
* do not have a present history of self-injury
* have tried fewer than four other treatment methods for self-injurious behavior
* if following their pre-treatment tests, they have medical conditions that would present them with undue risk for undergoing ECT.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Changes in Self-Injury Trauma Scale (SIT) across time | Baseline and weeks 7, 11, 6 months, and 12 months
  Self-Injury Trauma Scale (SIT). This scale allows differentiation and quantification of self-injury completed by the physician based on a complete medical assessment, location of injury, type of injury, number of injuries, and an estimate of severity.
  Scales include:
  * Number Index (NI) - Scores range from 0 (no current injuries) to 5 (17 or more current injuries)
  * Severity Index (SI) - Scores range from 0 (no current injuries) to 5 (maximum severity of current injuries)
  * Estimate of Current Risk - Scores range from Low (no current injuries or a lower level of injuries) to Moderate (any abrasion/laceration near the eyes OR any contusion except on the head) to High (any moderate contusion on the head OR any severe abrasion/laceration or contusion)

SECONDARY OUTCOMES:
Changes in Daily Diary Card across time | Baseline and weeks 2, 3, 4, 5, 6, 7, 11, 6 months, and 12 months
  A daily diary card used to record the number of self-injury episodes, the number of aggressive episodes, and the perceived severity of episodes per day.
Changes in Repetitive Behavior Scale-Revised (RBS-R) across time | Baseline and weeks 7, 11, 6 months, and 12 months
  The 43-item revised scale is specifically intended to assess the variety of repetitive behaviors in individuals with ASD, grouped into 6 categories: 1) stereotyped behavior, 2) self-injurious behavior, 3) compulsive behavior, 4) ritualistic behavior, 5) sameness behavior, and 6) restricted injurious behavior.
  All items are scored from 0 (behavior does not occur) to 1 (behavior occurs and is a mild problem) to 2 (behavior occurs and is a moderate problem) to 3 (behavior occurs and is a severe problem).
  Scale scores for the above 6 scales include:
  * Number of Subscale Items Endorsed: The total number of items in each scale rated 1, 2, or 3 (per scale)
  * Total Subscale Score: The sum of the ratings for all items in that scale (per scale)
  * Overall Number of Items Endorsed: The sum of all "Number of Subscale Items Endorsed" (combined scales Total score)
  * Overall Score: The sum of all "Total Subscale Scores" (combined scales Total score)
Changes in Aberrant Behavior Checklist (ABC) across time | Baseline and weeks 7, 11, 6 months, and 12 months
  A 58-item measure useful for evaluation inappropriate and maladaptive behavior with five subscales: 1) Irritability, Agitation, Crying; 2) Lethargy, Social Withdrawal; 3) Stereotypic Behavior; 4) Hyperactivity, Noncompliance; and 5) Inappropriate Speech.
  All items are scored from 0 (Not at all a problem) to 3 (the problem is severe in degree).
  Each of the 5 scales includes a sum of scores for items on that scale, ranging from [0] (no problem with this measure) to [12 to 48, depending on the scale] (severe problem with this measure).
Changes in ASD Diagnostic Checklist (ADC) across time | Baseline and weeks 7, 11, 6 months, and 12 months
  A 30-item instrument designed after the ADOS (Autism Diagnostic Observation Schedule), ADI-R (Autism Diagnostic Interview-Revised), and DSM-V (Diagnostic and Statistical Manual of Mental Disorders-V) criteria for autism, used to assess: 1) qualitative impairment in social interaction, 2) difficulties in communication, and 3) restricted, repetitive and stereotyped patterns of behavior.
  All items are scored "Yes" or "No".
  Scale scores are the sum of the number of "Yes" responses for each scale. Scores range from [0] (zero "Yes" responses equivalent to no ASD-related behaviors) to [6 to 14, depending on the scale] (all "Yes" responses equivalent to higher ASD-related behaviors).
  Total Score includes the sum of all items with a "Yes" response, ranging from 0 (no ASD-related behaviors) to 30 (higher ASD-related behaviors)

CONTACTS AND LOCATIONS:
Overall Officials: Shriti Patel, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tate BG, Baroff GS. Aversive control of self-injurious behavior in a psychotic boy. Behav Res Ther. 1966 Nov;4(4):281-7. doi: 10.1016/0005-7967(66)90024-6. No abstract available. PMID 5978683
- [Background] Iwata BA, Pace GM, Kissel RC, Nau PA, Farber JM. The Self-Injury Trauma (SIT) Scale: a method for quantifying surface tissue damage caused by self-injurious behavior. J Appl Behav Anal. 1990 Spring;23(1):99-110. doi: 10.1901/jaba.1990.23-99. PMID 2335488
- [Background] Wachtel LE, Dhossche DM. Self-injury in autism as an alternate sign of catatonia: implications for electroconvulsive therapy. Med Hypotheses. 2010 Jul;75(1):111-4. doi: 10.1016/j.mehy.2010.02.001. Epub 2010 Mar 3. PMID 20202760
- [Background] Dhossche DM, Carroll BT, Carroll TD. Is there a common neuronal basis for autism and catatonia? Int Rev Neurobiol. 2006;72:151-64. doi: 10.1016/S0074-7742(05)72009-2. PMID 16697296
- [Background] Dhossche DM. Autism as early expression of catatonia. Med Sci Monit. 2004 Mar;10(3):RA31-9. Epub 2004 Mar 1. PMID 14976444
- [Background] Chagnon YC. Shared susceptibility region on chromosome 15 between autism and catatonia. Int Rev Neurobiol. 2006;72:165-78. doi: 10.1016/S0074-7742(05)72010-9. PMID 16697297
- [Background] Hawkins JM, Archer KJ, Strakowski SM, Keck PE. Somatic treatment of catatonia. Int J Psychiatry Med. 1995;25(4):345-69. doi: 10.2190/X0FF-VU7G-QQP7-L5V7. PMID 8822386
- [Background] Rohland BM, Carroll BT, Jacoby RG. ECT in the treatment of the catatonic syndrome. J Affect Disord. 1993 Dec;29(4):255-61. doi: 10.1016/0165-0327(93)90015-c. PMID 8126312
- [Background] Haq AU, Ghaziuddin N. Maintenance electroconvulsive therapy for aggression and self-injurious behavior in two adolescents with autism and catatonia. J Neuropsychiatry Clin Neurosci. 2014 Winter;26(1):64-72. doi: 10.1176/appi.neuropsych.12110284. PMID 24515677
- [Background] Wachtel LE, Contrucci-Kuhn SA, Griffin M, Thompson A, Dhossche DM, Reti IM. ECT for self-injury in an autistic boy. Eur Child Adolesc Psychiatry. 2009 Jul;18(7):458-63. doi: 10.1007/s00787-009-0754-8. Epub 2009 Feb 5. PMID 19198918
- [Background] Wachtel LE, Griffin M, Reti IM. Electroconvulsive therapy in a man with autism experiencing severe depression, catatonia, and self-injury. J ECT. 2010 Mar;26(1):70-3. doi: 10.1097/YCT.0b013e3181a744ec. PMID 19483640
- [Background] Wachtel LE, Schuldt S, Ghaziuddin N, Shorter E. The potential role of electroconvulsive therapy in the 'Iron Triangle' of pediatric catatonia, autism, and psychosis. Acta Psychiatr Scand. 2013 Nov;128(5):408-9. doi: 10.1111/acps.12158. Epub 2013 Jun 17. No abstract available. PMID 23773168
- [Background] Zaw FK, Bates GD, Murali V, Bentham P. Catatonia, autism, and ECT. Dev Med Child Neurol. 1999 Dec;41(12):843-5. doi: 10.1017/s001216229900167x. PMID 10619284
- [Background] DeJong H, Bunton P, Hare DJ. A systematic review of interventions used to treat catatonic symptoms in people with autistic spectrum disorders. J Autism Dev Disord. 2014 Sep;44(9):2127-36. doi: 10.1007/s10803-014-2085-y. PMID 24643578
- [Background] Lam KS, Aman MG. The Repetitive Behavior Scale-Revised: independent validation in individuals with autism spectrum disorders. J Autism Dev Disord. 2007 May;37(5):855-66. doi: 10.1007/s10803-006-0213-z. PMID 17048092
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Dhossche DM, Reti IM, Wachtel LE. Catatonia and autism: a historical review, with implications for electroconvulsive therapy. J ECT. 2009 Mar;25(1):19-22. doi: 10.1097/YCT.0b013e3181957363. PMID 19190507
- [Background] Leyfer OT, Folstein SE, Bacalman S, Davis NO, Dinh E, Morgan J, Tager-Flusberg H, Lainhart JE. Comorbid psychiatric disorders in children with autism: interview development and rates of disorders. J Autism Dev Disord. 2006 Oct;36(7):849-61. doi: 10.1007/s10803-006-0123-0. PMID 16845581
- [Background] Mandell DS. Psychiatric hospitalization among children with autism spectrum disorders. J Autism Dev Disord. 2008 Jul;38(6):1059-65. doi: 10.1007/s10803-007-0481-2. Epub 2007 Nov 2. PMID 17975720
- [Background] Aman MG, Kasper W, Manos G, Mathew S, Marcus R, Owen R, Mankoski R. Line-item analysis of the Aberrant Behavior Checklist: results from two studies of aripiprazole in the treatment of irritability associated with autistic disorder. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):415-22. doi: 10.1089/cap.2009.0120. PMID 20973712
- [Background] Kaat AJ, Lecavalier L, Aman MG. Validity of the aberrant behavior checklist in children with autism spectrum disorder. J Autism Dev Disord. 2014 May;44(5):1103-16. doi: 10.1007/s10803-013-1970-0. PMID 24165702

DOCUMENTS (2):
  • Study Protocol (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03980366/Prot_000.pdf
  • Informed Consent Form (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03980366/ICF_001.pdf